CLINICAL TRIAL: NCT01729013
Title: Duration of Vitamin D Stores After Prolonged Vitamin D Substitution
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: Tromsø-Endo-2012-2
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: vitamin D; fat; biopsy
MeSH Terms: conditions — Obesity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and fat biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- subjects previously given placebo
- subjects previously given vitamin D

SUMMARY:
Ingested or skin produced vitamin D is either hydroxylated in the liver to 25-hydroxyvitamin D (25(OH)D), metabolized and excreted in the urine, or stored in adipose and other tissues. The capacity for vitamin D storage in adipose tissue is not known, nor the importance of such storage which may potentially be of vital importance when intake or solar exposure is limited. In the present study we will include 76 subjects who have participated in an intervention study with vitamin D (20.000 IU per week) versus placebo for the prevention of type 2 diabetes, and who have completed the study after 5 years or who have been excluded because of diagnosed type 2 diabetes or for other reasons. If vitamin D is stored to any extent in the body the subjects given 20.000 IU vitamin D per week for 2-5 years will have a considerable amount of stored vitamin D and accordingly, a slow decline in serum 25(OH)D during the following year without vitamin D substitution, which will be measured in the present study. If our hypothesis is correct, that vitamin D can be stored in significant amounts when the supply is abundant; current advice on vitamin D supplementation mainly during winter should be changed to "year around" in order to build up sufficient stores for the months without sufficient sun light.

ELIGIBILITY:
Inclusion Criteria:

* previously participated in a vitamin D study

Exclusion Criteria:

* pregnancy

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have previously participated in a vitamin D study
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
half-life of serum 25-hydroxyvitamin D | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: rolf jorde, professor, Principal Investigator — University of Tromso
Locations (1):
- University of Tromsø, Tromsø, Tromsø, Norway

REFERENCES:
- [Derived] Martinaityte I, Kamycheva E, Didriksen A, Jakobsen J, Jorde R. Vitamin D Stored in Fat Tissue During a 5-Year Intervention Affects Serum 25-Hydroxyvitamin D Levels the Following Year. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3731-3738. doi: 10.1210/jc.2017-01187. PMID 28973683